CLINICAL TRIAL: NCT06948188
Title: Identification of Subpopulations of Patients With Cholinergic Urticaria Based on the Results of Infrared Exposure
Brief Title: Identification of Subpopulations of Patients With Cholinergic Urticaria Based on Infrared Exposure Test Results.
Acronym: UCHOL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL_24_0383
Record Dates: First submitted 2025-03-31; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Cholinergic Urticaria
Keywords: cholinergic urticaria; urticaria; inducible urticaria; infrared radiation; dermatology, allergology; allergology
MeSH Terms: conditions — Urticaria

STUDY DESIGN:
Intervention Model Description: Single-center prospective interventional exploratory pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adult patients (> 18 years) with cholinergic urticaria (Experimental): Patient followed at Montpellier University Hospital with a diagnosis of cholinergic urticaria based on diagnostic criteria published in 2016 (Magerl et al): pruritic micropapules triggered by active or passive exposure to heat within 6 months following an exercise challenge test
  Interventions: Diagnostic Test: Infrared exposure test

INTERVENTIONS:
Diagnostic Test: Infrared exposure test — Patients will undergo a standardized infrared exposure test (this test is specifically for research purposes) to evaluate the occurrence of cholinergic urticaria reaction.
  IR exposure test with non-invasive core body temperature measurements, evaluate the occurrence of cholinergic urticaria up to 10 minutes after the end of the test, stop the test at the first clinical signs of urticaria.
  Desk lamp with infrared bulb, switched on 20cm vertically from the forearm posteriorly for 3 minutes. Reading up to 10 minutes after end of exposure test: diagnosis of cholinergic urticaria flare-up if presence of pruritic micropapules on erythematous background of trunk +/- limbs. Stop the test as soon as urticarial lesions appear.

SUMMARY:
This study aims to identify subpopulations of patients with cholinergic urticaria based on their sensitivity to infrared (IR) radiation exposure. Cholinergic urticaria is a chronic inducible urticaria triggered by increased body temperature. The study seeks to determine whether infrared exposure can induce symptoms in a subset of patients and whether these patients exhibit specific clinical or epidemiological characteristics.

DETAILED DESCRIPTION:
Cholinergic urticaria is characterized by small pruritic papules triggered by exercise, emotions, hot environments, or hot food and beverages. The pathophysiology remains unclear, but one hypothesis is that a central temperature increase plays a key role. A pilot study conducted at university hospital center (CHU) of Montpellier found that infrared exposure triggered symptoms in some patients with cholinergic urticaria. The infrared source was the same as that commonly used in photobiological tests.

The objective of this study is to identify the proportion of patients who develop cholinergic urticaria when exposed to infrared light. the investigators then aim to determine whether these patients have specific clinical or epidemiological characteristics that would allow them to be classified as a distinct subgroup of cholinergic urticaria and to assess whether sensitivity to infrared light is a prognostic marker of disease severity. Furthermore, measuring the core temperature of all patients during infrared light exposure will help determine whether patients sensitive to infrared light experience a greater increase in core temperature during the IR test. This would support the hypothesis that an increase in core temperature is responsible for triggering cholinergic urticaria flare-ups in this subgroup.

A better understanding of this condition and the identification of different subgroups could ultimately, with additional studies, allow for a personalized approach to patient management based on the cholinergic urticaria subgroup and each subgroup's sensitivity to different treatments.

ELIGIBILITY:
Inclusion criteria :

* Adults ≥ 18 years old
* Cholinergic urticaria diagnosed based on the diagnostic criteria published in 2016 (Magerl et al) : pruritic micropapules triggered by active or passive exposure to heat.
* Exercise test performed within the 6 months prior to inclusion.

Exclusion criteria :

* Patients on H1 antihistamines within 72 hours before infrared exposure test
* Patients on any other specific treatment for cholinergic urticaria within a period of 5 plasma half-lives before infrared exposure test
* Patients with exercise-induced anaphylaxis (diet-induced or not)
* Patients with severe forms of cholinergic urticaria: angioedema, respiratory manifestations or anaphylaxis
* Participants who have reached the maximum compensation amount for their participation in research studies.
* Lack of consent (adults, non-emancipated minors, individuals unable to express consent, research conducted in emergency situations, etc.).
* Not being affiliated with or a beneficiary of a French social security scheme.
* Protected adults (under guardianship, curatorship, or judicial protection).
* Individuals participating in another research study with an ongoing exclusion period.
* Subjects deprived of liberty (Art. L. 1121-6) (by judicial or administrative decision, or involuntary hospitalization).
* Pregnant or breastfeeding women.
* Subjects who cannot read and/or write.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2026-04-07 (Estimated); Study Completion 2026-04-07 (Estimated)

PRIMARY OUTCOMES:
Positive infrared test result | During the 3 minutes of exposure to infrared light and the following 10 minutes.
  the proportion (en percentage) of patients with cholinergic urticaria who develop urticarial lesions following infrared exposure.

SECONDARY OUTCOMES:
Comparison of age between patients with a positive and a negative infrared test | Baseline
  Epidemiological characteristics :
  age (year)
Comparison of age of onset of cholinergic urticaria, between patients with a positive and a negative infrared test | Baseline
  Epidemiological characteristics :
  age of onset of cholinergic urticaria (year)
Comparison of sex between patients with a positive and a negative infrared test | Baseline
  Epidemiological characteristics :
  sexe (male or female)
Comparison of history of atopy between patients with a positive and a negative infrared test | Baseline
  Epidemiological characteristics :
  history of atopy and/or angioedema and/or autoimmune diseases, (percentage between groups)
Comparison of associated chronic urticaria, between patients with a positive and a negative infrared test | Baseline
  Epidemiological characteristics :
  associated chronic urticaria,
Comparison of cholinergic urticaria activity score,between patients with a positive and a negative infrared test | Baseline
  Epidemiological characteristics :
  cholinergic urticaria activity score, CholUAS7
  Minimum Score: The minimum score for each item is 0. Maximum Score: The maximum score for each item is 3. For the weekly score (UAS7), which is the sum of daily scores over 7 days, the values range from 0 to 42, with higher values indicating greater disease activity.
Comparison of triggering factors between patients with a positive and a negative infrared test | Baseline
  Epidemiological characteristics :
  triggering factors of cholinergic urticaria (physical activity, heat exposure, consumption of hot or spicy foods, emotions),
Comparison of treatment effectiveness (between patients with a positive and a negative infrared test | Baseline
  Epidemiological characteristics :
  treatment effectiveness (antihistamines, omalizumab, and other treatments).
Comparison of time to onset of cholinergic urticaria (exercise) between patients with a positive and a negative infrared test | Baseline
  Clinical characteristics :
  time to onset of cholinergic urticaria during the exercise test on a stationary bike (seconds)
Comparison of time to onset of cholinergic urticaria (infrared) between patients with a positive and a negative infrared test | Baseline
  Clinical characteristics :
  time to onset of cholinergic urticaria during exposure to infrared light (if the test is positive),(seconds)
Comparison of maximum core temperature between patients with a positive and a negative infrared test | Baseline
  Clinical characteristics :
  non-invasive measurement of maximum core temperature during the infrared exposure test. (celcius)
Comparison of average core temperature between patients with a positive and a negative infrared test | Baseline
  Clinical characteristics :
  non-invasive measurement of average core temperature during the infrared exposure test. (celcius)

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie DU-THANH, MD, Principal Investigator — CHU de Montpellier
Locations (1):
- Chu de Montpellier, Montpellier, hérault, France

IPD SHARING:
Plan to Share IPD: Undecided